CLINICAL TRIAL: NCT04620876
Title: Bimodal and Coaxial High Resolution Ophtalmic Imaging
Acronym: AOSLO-OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P16-02; 2016-A00704-47 (Other: N° IDRCB)
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Retinitis Pigmentosa; Maculopathy, Age Related; Macular Dystrophy; Macular Edema; Retinal Detachment; Retinal Degeneration; Glaucoma; Vascular Inflammation; Hypertension; Stroke; Diabetes
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration; Macular Edema; Retinal Detachment; Retinal Degeneration; Glaucoma; Hypertension; Stroke; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bimodal and coaxial high resolution imaging of the retina (Experimental): Optical coherence tomography and Scanning laser ophthalmoscope system using adaptive optics (AO-SLO-OCT)
  Interventions: Other: Bimodal high resolution imaging of the retina

INTERVENTIONS:
Other: Bimodal high resolution imaging of the retina — The protocol consists of performing an Optical coherence tomography and Scanning laser ophthalmoscope system using adaptive optics (AO-SLO-OCT).The participant is asked to put his forehead against the temple supports and his chin on a chin rest. The subject will be asked to fix a test pattern in the form of a cross. The pattern is positioned according to the desired eccentricity with respect to the fovea. The actual acquisition lasts a few seconds, possibly repeated to cover the field of the desired eye. The acquisition protocol depends on the subjects, their pathology and the system used; the area examined will be modified on a case by case basis. The total duration of each exam can be estimated at less than half an hour, with frequent breaks.

SUMMARY:
The knowledge of the pathogenesis of retinal affections, a major cause of blindness, has greatly benefited from recent advances in retinal imaging. However, optical aberrations of the ocular media limit the resolution that can be achieved by current techniques.

The use of an adaptive optics system improves the resolution of ophthalmoscopes by several orders of magnitude, allowing the visualization of many retinal microstructures: photoreceptors, vessels, bundles of nerve fibers.

Recently, the development of the coupling of the two main imaging techniques, the Adaptive Optics Ophthalmoscope with Optical Coherence Tomography, enables unparalleled three-dimensional in vivo cell-scale imaging, while remaining comfortable for the patients.

The purpose of this project is to evaluate the performance of this system for imaging micrometric retinal structures.

DETAILED DESCRIPTION:
The goal of the project is the capture and analysis of images with AOSLO system, in order to evaluate the performance of this system compared to OCT imaging devices and existing Adaptive Optics used at National Hospital of Ophthalmology.

ELIGIBILITY:
Inclusion Criteria:

* People over 18
* Patient with a pathology affecting the eye or healthy volunteer
* Participant who signed the consent
* Beneficiaries of the health insurance

Exclusion Criteria

* Patients with a history of photosensitivity.
* Patients who have just received a photodynamic therapy treatment
* Patients taking drugs with photosensitivity as a side effect.
* Persons with pacemakers or other implanted electronic medical device
* Patients with viral conjunctivitis or any other infectious disease.
* Patients with skin lesions on the neck or forehead
* Patients at high risk of damage from optical radiation, such as aphakic patients, or patients with decreased sensitivity to light due to fundus disease.
* Participant unable to be followed throughout the study
* Advanced cataract or severe opacities in the anterior segment of the eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Visualization and image analysis of a structure of interest | From date of inclusion until the date of last documented progression , assessed up to 5 years
  The visualization of the structure of interest in at least one area of the image will be considered the main criterion of success.

CONTACTS AND LOCATIONS:
Overall Officials: Michel PAQUES, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France